CLINICAL TRIAL: NCT02065128
Title: The Efficacy of Capsaicin Sensitivity Testing in Patients With Irritable Larynx Syndrome
Status: Withdrawn | Type: Observational
Why Stopped: Logistical challenges with research pharmacy prevented the dilution of the capsaicin. No participants were ever recruited, enrolled, or approached.
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 14-005
Record Dates: First submitted 2014-02-11; First posted 2014-02-17 (Estimated); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Cough; Larynx
MeSH Terms: conditions — Cough; Laryngeal Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy Volunteers: Capsaicin cough challenge test. The ILS participants will be asked to attend two study visits at the pulmonary function laboratory at SMH; one before behavioural therapy and one after. The healthy volunteers will be asked to attend one study visit. At each of these study visits, the ILS participants will complete the Leicester Cough Questionnaire (LCQ) (Appendix B) and the Dyspnea Index (DI) Questionnaire (Appendix C). The LCQ is a valid assessment tool for evaluating the impact of cough on QoL.19 The DI is a short, validated questionnaire used to quantify a patient's symptoms of dyspnea.20 Following completion of the questionnaires, participants will complete a capsaicin cough challenge test, which is discussed in the following section.
  Interventions: Other: Capsaicin cough challenge test
- Irritable Larynx Syndrome Patients: Capsaicin cough challenge test. The ILS participants will be asked to attend two study visits at the pulmonary function laboratory at SMH; one before behavioural therapy and one after. The healthy volunteers will be asked to attend one study visit. At each of these study visits, the ILS participants will complete the Leicester Cough Questionnaire (LCQ) (Appendix B) and the Dyspnea Index (DI) Questionnaire (Appendix C). The LCQ is a valid assessment tool for evaluating the impact of cough on QoL.19 The DI is a short, validated questionnaire used to quantify a patient's symptoms of dyspnea.20 Following completion of the questionnaires, participants will complete a capsaicin cough challenge test, which is discussed in the following section.

INTERVENTIONS:
Other: Capsaicin cough challenge test — The capsaicin cough challenge testing will be conducted in the pulmonary function laboratory at SMH by a pulmonary function technologist. The test involves having the participant inhale increasing concentrations of capsaicin solutions and assessing their response. The tidal breathing method and solution preparation presented by Nejla, et al. 12 will be used to conduct this testing. The tidal breathing method is preferred to the alternative dosimeter method as it produces similar results with lower capsaicin concentrations thereby resulting in less throat irritation for the participant. The technique is detailed in the following sections.
  Groups: Healthy Volunteers

SUMMARY:
Irritable larynx syndrome (ILS) is a hyperkinetic laryngeal dysfunction that is characterized by a persistent cough, voice changes, or breathing difficulties, which are often triggered by an irritant. Diagnosis of ILS is difficult and typically made via a thorough review of the clinical history and, occasionally, the patient's reaction to an odor-provocation test. Standard treatment for ILS is behavioural therapy with a speech language pathologist (SLP), which provides symptom improvement for most patients. However, currently, there are no objective measures of the upper airway hyper-responsiveness in this condition to assist in diagnosing and monitoring disease severity.

Since the cough is irritant-based, it is anticipated that patients with ILS will have a hypersensitivity to the irritant capsaicin. Capsaicin is the active component of chili peppers and is what makes them hot. The capsaicin cough challenge is a well recognized test that involves inhaling different concentrations of capsaicin solutions to determine a cough reflex sensitivity.

The purpose of this research study is to confirm that ILS patients have a hypersensitivity to capsaicin compared to healthy volunteers. If a hypersensitivity is observed in ILS patients, the second objective of this study will be to see if behavioural therapy improves the cough reflex sensitivity in this patient population.

DETAILED DESCRIPTION:
The proposed study has two purposes; the first is to utilize capsaicin cough challenge to demonstrate an increased efferent receptor sensitivity level in ILS subjects as compared to a control group. The second is to determine if there is an objective change in capsaicin cough challenge results after behavioral therapy, and whether it correlates to the subjective improvement. Self-reporting measures include two validated cough quality of life (QoL) questionnaires collected at the same intervals as the capsaicin testing.

ELIGIBILITY:
ILS Participants:

Inclusion Criteria:

* Diagnosis of ILS as per the St Michael's voice clinic consultation
* Methacholine test performed
* Negative/borderline result for methacholine test and/or negative/incomplete response for asthma treatment
* Negative test result for gastroesophageal reflux or negative/incomplete response to reflux treatment
* Allergy test has been completed with negative result or does not account for all symptoms
* Agreed to behavioural therapy in SMH Voice Disorders Clinic

Exclusion Criteria:

* Active smoker
* Active respiratory disease (e.g., COPD, pulmonary fibrosis, lung malignancy.)
* Taking an ACE inhibitor
* Pregnant and/or breastfeeding
* Impaired liver and/or renal function
* Neurological disorder
* Psychiatric condition (outside of depression or anxiety)

Healthy Volunteers:

Exclusion Criteria:

* Active smoker
* Active respiratory disease (e.g. COPD, asthma)
* ILS diagnosis
* Chronic cough diagnosis
* Known hypersensitivity to capsaicin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ILS Patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
cough reflex sensitivity | measured before and after behavioural therapy for ILS participants (approximately 5 month time frame); measured once for healthy volunteers
  measured via the capsaicin cough challenge test

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Anderson, MD, FRCS(C), Principal Investigator — Chief, Department of Otolaryngology - Head and Neck Surgery
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada